CLINICAL TRIAL: NCT07004036
Title: The Effects Of Occupation-Based Self-Regulation Program On Sensory Processing, Executive Functions and Occupational Performance In Preschool Children With Screen Addiction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Yasin Tekeci, PhD Lecturer, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023/84-2023080
Record Dates: First submitted 2025-05-18; First posted 2025-06-04 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Screen Time Exposure
Keywords: Screen Time Exposure; Executive Function; Self-control; Sensory Processing
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Intervention Model Description: One group will receive one-time family training on screen addiction and its harms, while the other group will receive a self-regulation intervention program in addition to family training.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): All 20 children participating in the study are individuals who have more than 2 hours of screen time per day. The individuals in the study do not have any known diagnosis that affects their self-regulation skills. Both their families and themselves are participating in the study voluntarily. They are randomly divided into two groups of 10 people. Each arm consists of 10 individuals. This is an intervention program that will be applied to the individuals in this arm for 8 weeks regarding self-regulation skills. During these eight weeks, one session per week will be applied in groups and one session will be applied individually. The intervention will include sensory processing skills and executive function skills. In addition, awareness training was provided to the families of the participants in this arm about the effects and harms of screen addiction.
  Interventions: Behavioral: Occupation-based Self-Regulation Intervention Program
- Control Group (Other): All 20 children participating in the study were individuals who had more than 2 hours of screen time per day. The individuals in the study did not have any known diagnosis that affected their self-regulation skills. Both their families and themselves participated in the study voluntarily. They were randomly divided into two groups of 10 people. Each arm consisted of 10 individuals. Awareness training was provided to the families of the participants in this arm about the effects and harms of screen addiction.
  Interventions: Behavioral: Family Awareness Training

INTERVENTIONS:
Behavioral: Occupation-based Self-Regulation Intervention Program — The intervention includes both group and individual applications. It has a large occupation/activity pool that can be selected in a person-centered manner. The activities are focused on supporting and developing the areas of influence in the sensory processing skills of individuals or the areas in executive functions, and providing occupations that will replace the screen and shape life in children for the screen abuse. It shapes the will, habits and routines necessary for the child to prefer alternative activities instead of the screen. For this purpose, an intervention program has been shaped to ensure that the child gains in the areas of daily life activities, productivity activities and leisure activities with the right developing skills, the child's wishes, the family's wishes, social expectations. As far as we know, it is the first flood regulation intervention program applied to children with screen addiction from an occupational therapy perspective.
  Arms: Intervention Group
Behavioral: Family Awareness Training — Family awareness training on the harms of screen addiction and prolonged exposure to the screen, as a one-time event.
  Arms: Control Group

SUMMARY:
The purpose of this interventional study was to measure the effectiveness of a self-regulation program for screen addiction in preschool children aged 4-5 years. The main questions it aimed to answer were:

Does a self-regulation intervention program reduce screen addiction in preschool children? Does a self-regulation intervention program improve self-regulation skills in preschool children? Does a self-regulation intervention program improve sensory processing skills in preschool children? Does a self-regulation intervention program improve reading performance in preschool children?

DETAILED DESCRIPTION:
Time spent using screen-based media devices is present in every aspect of the lives of twenty-first-century children and adults. Rapid technological advances and the marketing of portable screen-based devices such as smartphones and tablets to consumers around the world have changed the way and duration of people interacting with electronic media. As our society becomes more technologically dependent, the health effects of high levels of sedentary screen time, especially among children and adolescents, need to be given more attention. Defined as time spent watching television, DVDs, or videos or playing computer or video games, screen time has been linked to serious health outcomes in children, including impaired language acquisition, violent behavior, tobacco smoking, and obesity. In 2001, the American Academy of Pediatrics recommended that children under 2 should not spend time in front of a screen at all, limited it to one hour per day from age 2 to age 5, and recommended a two-hour limit for daily screen time for non-school and/or non-work activities after age 5, and today offers a general recommendation to limit screen time. Despite these recommendations, the time spent in front of screens has been increasing day by day, while the age of use has decreased from 4 years to 4 months since the 1970s.

The term "screen addiction" is increasingly used to describe the increasing number of children who engage in various screen activities in a dependent and problematic manner. The concept and diagnostic criteria are derived from criteria for pathological gambling and substance-related addiction and are generally based on the amount of time spent on a screen activity, such as playing the computer, and the extent to which it compromises the individual's overall functioning. Similar to other addictions, the diagnostic criteria include preoccupation, withdrawal symptoms, increased tolerance, failure to reduce or stop screen activities, loss of other interests, continuation despite negative consequences, lying about the extent of use, and use to escape negative moods.

The main neurological interest has focused on the problematic use of internet and computer games. However, although there is currently a degree of interchangeability and overlap between some diagnostic and diagnostic terms, the lack of standardization in concepts and terminology is considered a major obstacle to advancing this area of research and treatment, and steps are being taken to achieve greater consensus on terminology. Therefore, addictions such as internet addiction disorder, internet gaming disorder, problematic internet use, compulsive internet use, pathological video game use, video game addiction, pathological technology use, online gaming disorder, mobile phone addiction, social networking addiction, Facebook addiction, internet pornography addiction are all considered screen addiction disorders. There is a steady increase in young people's digital media consumption in most Western and some Far Eastern countries. In 2011, 52% of children aged 0-8 had access to a mobile device. This access increased to 75% by 2013 (8). In 1999, the average screen time of 8-18 year olds was 6.21 hours per day and increased to 7.38 hours in 2009. A self-reported study of screen time habits shows that British children and adolescents (8-18) spend an average of 4 hours and 45 minutes per day in front of a screen, either as a main activity or when engaged in other activities. Furthermore, the results from the same study show a significant increase in screen time among British children from 2010 to 2015. In most age groups in North America, there has been a significant increase in computer use in leisure time from 2001 to 2016. According to a 2018 survey of 3660 school children in Denmark, 24% of boys and 19% of girls aged 13-15 watch at least four hours of movies, TV series, YouTube films or entertainment programs per weekday. A study of more than 2,000 U.S. children ages 8 to 18 found that 21% typically watched more than 16 hours of media content in a 24-hour period, 63% watched 3 to 16 hours, and only 17% watched less than 3 hours. In addition, the International Child Accelerometer Database found that in a sample of 11,434 children ages 4 to 17, at least two-thirds had more than 2 hours of screen time. These findings suggest that an alarming number of children and adolescents are engaging in excessive sedentary screen time, leading to a range of adverse health outcomes.

Preschool children who spend 1 hour or more per day in early childhood and 2 hours or more per day after the age of 5 may experience a number of negative problems related to child health and well-being. Many problems such as unhealthy eating patterns, obesity, poor sleep quality, orthopedic problems, cardiovascular diseases, increased emotion dysregulation, decreased prosocial behaviors, increased inattention and hyperactivity, lower language skills, executive dysfunction, cognitive problems, and disruptions in the parent-child relationship, including reading books together, have been associated with increased screen time. However, childhood is a period when there are significantly greater changes in the anatomical structure and connectivity of the brain. It has been suggested that screen addiction disorder, and even intensive exposure to screens such as intensive video game play during childhood, may lead to neuroadaptations and structural changes in neural regions associated with addiction. In a study of 248 healthy children aged 5-17, Takeuchi et al. They reported significant correlations between average daily video game playing hours over a 3-year period and microstructural changes that reflected a decrease in tissue density. These changes were uniquely susceptible to neural plasticity, particularly within the dopaminergic system. Consequently, increased video gaming is directly and indirectly associated with delayed microstructural development in large brain regions. Conditions in which children play video games for long periods of time may lead to adverse neurocognitive development. These brain regions are often the same brain regions implicated in gambling disorders and substance abuse studies. The development and maintenance of video game addiction is increasingly viewed as a maladaptive interaction between neurological structures and functions underlying important components of addiction: reward, pleasure, craving, reinforcement, learning, memory, impaired executive functions, inhibitory control, decision making, and emotion management. Much of the neurological research on video game addiction has focused on dysfunctional interactions between neurological structures involved in executive control and reward seeking. Structural differences between subjects with and without SAD have been reported in additional brain regions, such as prefrontal and limbic structures in both gray and white matter. Functional brain correlates of SAD are also found in the prefrontal cortex and limbic structures. The typical features of impaired executive function and inhibitory control in addiction are related to low functional connectivity in fronto-striatal circuits. Changes in dopaminergic systems related to reinforcement/reward processing have also been suggested. Recent whole-brain functional connectivity analyses in SAD subjects have indicated that there are predominantly impaired connections in frontal areas, representing changes underlying different aspects of cognitive control. Interestingly, impairments similar to clinical cases have been shown in the preclinical stages of Internet addiction. However, the authors state that 'the interregional connections associated with Internet addiction tendencies replicate those frequently seen in the substance addiction literature'. In the study conducted by Wang et al., compared to the control group, subjects with internet gaming disorder had increased functional connectivity problems in the prefrontal cortex, left posterior cingulate cortex, right amygdala and bilateral lingual gyrus, and sensory-motor brain networks, along with functional connectivity disorders including impaired executive control and emotional management.

Since sensory-perceptual abnormalities are manifestations of disorders in the interactions of the neocortex, basal ganglia, and cerebellum, they are likely to coexist with abnormalities in motor function, cognitive and communication deficits, and social functioning. This is because sensory processing abnormalities are subtle indicators of deficits in "executive control," broadly defined. This is because sensory processing skills are more apparent in the developing brain, where they can be diagnosed earlier than more complex executive control can be measured, and executive control can be measured later when conditions are favorable. The development of working memory functions depends on inhibitory control. In the absence of inhibitory capacity to sustain focused attention, thought-guided behavior is inhibited. Deficits in cognitive abilities, emotional control, academic skill sets, and even communication and social competence can all be predicted based on the regions and extent of pathology in brain systems that mediate choice and regulation. In this context, early detection of hypo and/or hypersensitivity and responsiveness may enable the development of treatment approaches that increase compliance in various functional areas.

In a study conducted to define the relationship between the time children spend in front of the screen and sensory processing skills, a significant and negative relationship was found specifically between visual, tactile, body awareness, balance, planning and general sensory processing skills. It has been stated that in connection with the increased screen exposure time of children at an early age, there are problems such as "decreased cognitive abilities, poor school performance, slowed growth, development of addictive behavior, poor sleep patterns and increased obesity levels" which can be said to be related to sensory processing problems.

If the sensory processing system does not provide reliable information, sensory processing disorder may occur. In this case, the person's organizational, motor, attention, self-care, auditory and visual skills are negatively affected and the individual may not feel safe.

Although the development of executive functions has its roots in infancy, it begins to develop at approximately 4 years of age. Executive functions such as task persistence, impulse control, emotion regulation, and creativity and cognitive flexibility are affected by child-led play as well as positive parenting. Recent studies have shown associations between media use in childhood and poorer executive function. These studies suggest that earlier age at which media use begins and higher cumulative hours of media use are important independent predictors of poor executive function. This association has been attributed to the stimulating and fast-paced content of some children's schedules and the displacement of other enriching activities or the time when the brain is not functionally engaged. Media multitasking, which is associated with executive function deficits in young adults, has now been documented in children as young as 4 years old.

Screen addiction disorder, which has been shown to have executive function deficits and sensory processing deficits, also has speech organization problems in children with screen addiction-intense screen time.

Preschool children have cognitive developmental problems or sensory processing problems, along with accompanying problems in participation in activities of daily living, leisure time, and play. Studies have shown that activity participation and activity performance are affected in children with sensory processing problems, cognitive problems, especially executive dysfunctions, attention deficit and hyperactivity disorder, or various disorders such as autism spectrum disorder. Occupational performance is a dynamic process that covers the entirety of an individual's daily life activities and is affected by many factors such as physical, cognitive, emotional, environmental and social patterns. Studies have suggested that the situation defined as nomophobia, which is defined as the fear of being away from a mobile phone, has a negative effect on ADL because it causes problems in cognitive, emotional, physical and social functions. The concept of self-regulation, which is extremely important for children to be able to regulate their cognitions, emotions and behaviors on their own, to be ready for school, and to be successful in school and in their future lives, is described in the literature as a broad term that includes planning and executive skills (especially working memory, cognitive flexibility and inhibitory control) as top-down and regulation of reactive impulses as bottom-up.

ELIGIBILITY:
Inclusion Criteria:

* Children between 48-59 months of age
* Who do not have any additional diagnosis
* Spend 2 hours or more on screens per day and
* Attend kindergarten will be included.

Exclusion Criteria:

* Have any diagnosed disorder that may cause sensory processing disorder or executive function disorder,
* Have any diagnosed disorder that may lead to limitation of occupational performance, or
* Individuals who have not attended kindergarten will not be included in the study.

Ages: 48 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Screen Time | The average daily screen time for one week at the beginning of the study and the average daily screen time for one week at the end will be measured.
  The average daily screen time for one week at the beginning of the study and the average daily screen time for one week at the end will be measured.
Sensory Processing | Both assessments will take 15 minutes each, one at the beginning of the study, the day before the intervention, and one at the end of the study, the day after the intervention.
  The Dunn Sensory Profile was developed to assess responses in children to a variety of common sensory experiences. Parents are asked to rate the frequency of responses in their children to 125 common experiences using a Likert scale format. These questions and responses are divided into eight categories: Auditory, Visual, Activity Level, Taste/Smell, Body Position, Movement, Touch, and Emotional/Social. The sensory profile was deemed appropriate for children ages 3-10 and was standardized on 1,200 children with and without disabilities. Content and construct validity have been established. Responses are summarized in six sensory processing domains (Auditory Processing, Visual Processing, Vestibular Processing, Tactile Processing, Multisensory Processing, Oral Sensory Processing), five modulation processes, and three behavioral and emotional responses domains. The validity and reliability studies of the scale in Turkish.
Executive Function/Self Regulation | Both assessments will take 30 minutes each, one at the beginning of the study, the day before the intervention, and one at the end of the study, the day after the intervention.
  The scale consists of 3 levels of applications. At the first level, the child is asked to touch his feet when he is told to "touch his head" and to touch his head when he is told to "touch his feet". If he is successful at this level, he is asked to touch his shoulders when he is told to "touch his knee" and to touch his knees when he is told to "touch his shoulder". If he is successful at this level, he is asked to touch his knees when he is told to "touch his head", to touch his shoulders when he is told to "touch his feet", to touch his feet when he is told to "touch his shoulder" and to touch his head when he is told to "touch his knees". If he can do the given command without any mistakes, he is given 2 points, if he is oriented towards the wrong and does it correctly, he is given 1 point and if he gives the wrong answer, he is given 0 points. A total score of 0-60 is given with 10 applications at each level. As the score increases, the self-regulation score will increase.
Occupational Performance | Both assessments will take 10 minutes each, one at the beginning of the study, the day before the intervention, and one at the end of the study, the day after the intervention.
  The Canadian Occupational Performance Measure (COPM) is a general questionnaire based on a semistructured interview. The semistructured design allows individuals to identify important occupations that they have difficulty performing. COPM is derived from the Canadian Activity Performance Model, which defines occupational performance as the ability to organize, select, and perform meaningful occupations that are culturally defined and age-appropriate for taking care of oneself, enjoying life, building the economic fabric of society, and contributing to the social world. The fifth version of the COPM was published in 2014 and its Turkish adaptation has been made.
Problematic Media Use | Both assessments will take 5 minutes each, one at the beginning of the study, the day before the intervention, and one at the end of the study, the day after the intervention.
  It was developed to determine problematic media use in children between the ages of 4 and 11. The items of the scale were created by taking into account the Internet Gaming Disorder criteria expressed in DSM V. The scale consists of a 27-item form. The scale is Likert-type and each item is scored between 1 (never) and 5 (always). The total score obtained from the Problematic Media Use Scale is calculated by averaging the scores obtained from all items. High scores obtained from the scale indicate problematic use. While the scale, which is filled out by parents considering the child's behavior, does not provide information on the problematic use of a specific media tool, it tries to determine the problematic use of visual media tools (such as phones, tablets, computers, televisions) in general, in other words, screen addiction.
Occupational Profile | Both assessments will take 10 minutes each, one at the beginning of the study, the day before the intervention, and one at the end of the study, the day after the intervention.
  This assessment tool comprises 25 items organized into six sections. The initial five sections (volition, habituation, communication & interaction skills, process skills, motor skills) evaluate the child's personal attributes and their influence on participation and performance in various activities. The final section investigates the impact of the environment on the child's capacity to engage in and perform these activities.
  A four-point ordinal scale is employed for scoring individual items, using the following codes:
  F = Facilitates A = Allows I = Inhibits R = Restricts participation
  Numerical values are assigned to each code, ranging from 4 to 0. Specifically, 'F' is assigned a value of 4, 'A' is 3, 'I' is 2, and 'R' is 1.
  The item scores are summed, yielding a maximum total score of 100 for the entire assessment. The minimum score is 25.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Argumosa-Villar L, Boada-Grau J, Vigil-Colet A. Exploratory investigation of theoretical predictors of nomophobia using the Mobile Phone Involvement Questionnaire (MPIQ). J Adolesc. 2017 Apr;56:127-135. doi: 10.1016/j.adolescence.2017.02.003. Epub 2017 Feb 21. PMID 28231484
- [Background] Carswell A, McColl MA, Baptiste S, Law M, Polatajko H, Pollock N. The Canadian Occupational Performance Measure: a research and clinical literature review. Can J Occup Ther. 2004 Oct;71(4):210-22. doi: 10.1177/000841740407100406. PMID 15586853
- [Background] Wennberg B, Janeslatt G, Gustafsson PA, Kjellberg A. Occupational performance goals and outcomes of time-related interventions for children with ADHD. Scand J Occup Ther. 2021 Feb;28(2):158-170. doi: 10.1080/11038128.2020.1820570. Epub 2020 Sep 21. PMID 32955952
- [Background] Mathews, S. B., Mozolic-Staunton, B., Jefford, E., & Salehi, N. (2020). Canadian Occupational Performance Measure and early intervention: A scoping review. Journal of Occupational Therapy, Schools, & Early Intervention, 13(4), 353-373.
- [Background] Dadson P, Brown T, Stagnitti K. Relationship between screen-time and hand function, play and sensory processing in children without disabilities aged 4-7 years: A exploratory study. Aust Occup Ther J. 2020 Aug;67(4):297-308. doi: 10.1111/1440-1630.12650. Epub 2020 Jan 30. PMID 32003027
- [Background] Koziol LF, Budding DE, Chidekel D. Sensory integration, sensory processing, and sensory modulation disorders: putative functional neuroanatomic underpinnings. Cerebellum. 2011 Dec;10(4):770-92. doi: 10.1007/s12311-011-0288-8. PMID 21630084
- [Background] Wang L, Wu L, Lin X, Zhang Y, Zhou H, Du X, Dong G. Altered brain functional networks in people with Internet gaming disorder: Evidence from resting-state fMRI. Psychiatry Res Neuroimaging. 2016 Aug 30;254:156-63. doi: 10.1016/j.pscychresns.2016.07.001. Epub 2016 Jul 6. PMID 27447451
- [Background] Brand M, Young KS, Laier C, Wolfling K, Potenza MN. Integrating psychological and neurobiological considerations regarding the development and maintenance of specific Internet-use disorders: An Interaction of Person-Affect-Cognition-Execution (I-PACE) model. Neurosci Biobehav Rev. 2016 Dec;71:252-266. doi: 10.1016/j.neubiorev.2016.08.033. Epub 2016 Aug 30. PMID 27590829
- [Background] Takeuchi H, Taki Y, Hashizume H, Asano K, Asano M, Sassa Y, Yokota S, Kotozaki Y, Nouchi R, Kawashima R. Impact of videogame play on the brain's microstructural properties: cross-sectional and longitudinal analyses. Mol Psychiatry. 2016 Dec;21(12):1781-1789. doi: 10.1038/mp.2015.193. Epub 2016 Jan 5. PMID 26728566
- [Background] Atkin AJ, Sharp SJ, Corder K, van Sluijs EM; International Children's Accelerometry Database (ICAD) Collaborators. Prevalence and correlates of screen time in youth: an international perspective. Am J Prev Med. 2014 Dec;47(6):803-7. doi: 10.1016/j.amepre.2014.07.043. Epub 2014 Sep 16. PMID 25241193
- [Background] Rasmussen M, Damsgaard MT, Morgen CS, Kierkegaard L, Toftager M, Rosenwein SV, Krolner RF, Due P, Holstein BE. Trends in social inequality in overweight and obesity among adolescents in Denmark 1998-2018. Int J Public Health. 2020 Jun;65(5):607-616. doi: 10.1007/s00038-020-01342-1. Epub 2020 Feb 20. PMID 32076738
- [Background] Yang L, Cao C, Kantor ED, Nguyen LH, Zheng X, Park Y, Giovannucci EL, Matthews CE, Colditz GA, Cao Y. Trends in Sedentary Behavior Among the US Population, 2001-2016. JAMA. 2019 Apr 23;321(16):1587-1597. doi: 10.1001/jama.2019.3636. PMID 31012934
- [Background] Magee CA, Lee JK, Vella SA. Bidirectional relationships between sleep duration and screen time in early childhood. JAMA Pediatr. 2014 May;168(5):465-70. doi: 10.1001/jamapediatrics.2013.4183. PMID 24589672
- [Background] Reid Chassiakos YL, Radesky J, Christakis D, Moreno MA, Cross C; COUNCIL ON COMMUNICATIONS AND MEDIA. Children and Adolescents and Digital Media. Pediatrics. 2016 Nov;138(5):e20162593. doi: 10.1542/peds.2016-2593. PMID 27940795
- [Background] Radesky JS, Christakis DA. Increased Screen Time: Implications for Early Childhood Development and Behavior. Pediatr Clin North Am. 2016 Oct;63(5):827-39. doi: 10.1016/j.pcl.2016.06.006. PMID 27565361
- [Background] American Academy of Pediatrics. Committee on Public Education. American Academy of Pediatrics: Children, adolescents, and television. Pediatrics. 2001 Feb;107(2):423-6. doi: 10.1542/peds.107.2.423. PMID 11158483
- [Background] Lissak G. Adverse physiological and psychological effects of screen time on children and adolescents: Literature review and case study. Environ Res. 2018 Jul;164:149-157. doi: 10.1016/j.envres.2018.01.015. Epub 2018 Feb 27. PMID 29499467
- [Background] Rasmussen MGB, Pedersen J, Olesen LG, Brage S, Klakk H, Kristensen PL, Brond JC, Grontved A. Short-term efficacy of reducing screen media use on physical activity, sleep, and physiological stress in families with children aged 4-14: study protocol for the SCREENS randomized controlled trial. BMC Public Health. 2020 Mar 23;20(1):380. doi: 10.1186/s12889-020-8458-6. PMID 32293374
- [Background] Torpil B, Ekici Caglar G, Bumin G, Pekcetin S. Validity and Reliability of the Turkish Canadian Occupational Performance Measure (COPM-TR) for People with Multiple Sclerosis. Occup Ther Health Care. 2021 Jul;35(3):306-317. doi: 10.1080/07380577.2021.1933673. Epub 2021 Jun 14. PMID 34126836
- [Background] Bowyer, P., Lee, J., Kramer, J., Taylor, R.R., Kielhofner, G. (2012). Determining the clinical utility of the Short Child Occupational Profile (SCOPE). British Journal of Occupational, 75(1), 19.
- [Background] Domoff SE, Harrison K, Gearhardt AN, Gentile DA, Lumeng JC, Miller AL. Development and Validation of the Problematic Media Use Measure: A Parent Report Measure of Screen Media "Addiction" in Children. Psychol Pop Media Cult. 2019 Jan;8(1):2-11. doi: 10.1037/ppm0000163. Epub 2017 Nov 16. PMID 30873299
- [Background] McClelland MM, Cameron CE, Duncan R, Bowles RP, Acock AC, Miao A, Pratt ME. Predictors of early growth in academic achievement: the head-toes-knees-shoulders task. Front Psychol. 2014 Jun 17;5:599. doi: 10.3389/fpsyg.2014.00599. eCollection 2014. PMID 25071619
- [Background] Kayihan H, Akel BS, Salar S, Huri M, Karahan S, Turker D, Korkem D. DEVELOPMENT OF A TURKISH VERSION OF THE SENSORY PROFILE: TRANSLATION, CROSS-CULTURAL ADAPTATION, AND PSYCHOMETRIC VALIDATION. Percept Mot Skills. 2015 Jun;120(3):971-86. doi: 10.2466/08.27.PMS.120v17x8. Epub 2015 Jun 9. PMID 26057421
- [Background] Kashefimehr B, Kayihan H, Huri M. The Effect of Sensory Integration Therapy on Occupational Performance in Children With Autism. OTJR (Thorofare N J). 2018 Apr;38(2):75-83. doi: 10.1177/1539449217743456. Epub 2017 Dec 27. PMID 29281930
- [Background] Bowyer PL, Kramer J, Kielhofner G, Maziero-Barbosa V, Girolami G. Measurement properties of the Short Child Occupational Profile (SCOPE). Phys Occup Ther Pediatr. 2007;27(4):67-85. PMID 18032150